CLINICAL TRIAL: NCT00474461
Title: Myocardial Regeneration Using Cardiac Stem Cells Harvested From Right Atrial Appendages in Patients With Ischemic Cardiomyopathy.
Brief Title: Cardiac Stem Cell Infusion in Patients With Ischemic CardiOmyopathy (SCIPIO)
Acronym: SCIPIO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Brigham and Women's Hospital (Other); Jewish Hospital and St. Mary's Healthcare (Other)
Responsible Party: Principal Investigator, Roberto Bolli, Chief of the Division of Cardiovascular Medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOIC070833
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Congestive Heart Failure
Keywords: coronary artery disease; Heart Attack; Heart failure; Cardiac Stem Cells; Coronary Artery Bypass
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Patients in this arm received intracoronary expanded autologous c-kit positive cardiac stem cells.
  Interventions: Biological: Treatment group
- Control group (No Intervention): Patients in this arm did not receive any intervention.

INTERVENTIONS:
Biological: Treatment group — Intracoronary injection of cardiac stem cells
  Other Names: Intracoronary Injection (cardiac stem cell therapy)
  Arms: Treatment group

SUMMARY:
The purpose of this study is to investigate the safety of intracoronary cardiac stem cells (CSCs) therapy in humans. Currently, there is no effective intervention to regenerate (regrow) dead heart muscle after a heart attack.

The central hypothesis is that CSCs infused into nonviable myocardial segments will regenerate infarcted myocardium by differentiating into cardiomyocytes and other cell types. According to our hypothesis, CSC infusion regenerates myocardium with consequent improvement in contractile function of the heart and general clinical status.

DETAILED DESCRIPTION:
This will be a randomized, open-label study involving 20 patients and 20 controls. This study will be done as a collaborative project between Brigham Women's Hospital and The University of Louisville. This study is a phase I trial assessing the safety and feasibility of intracoronary autologous CSC [harvested from the right atrial appendage (RAA)] transplantation in patients with ischemic cardiomyopathy. The study will be conducted in two stages: Stage A, in which the investigators will obtain an initial assessment of safety and feasibility, and stage B, in which the investigators will adopt a block randomization strategy that will enable us to assess the feasibility of conducting a subsequent, randomized phase II trials. While the investigators also hope to have an estimate of efficacy, this focus will be the specific aim of future phase II trials. All patients who are undergoing on-pump CABG will be screened twice. The initial screening will be done to determine the preliminary eligibility (before-CABG screening) of patients for the study. If the patients satisfy the preliminary eligibility criteria stated below, the right atrial appendage, which is routinely resected during all on-pump bypass surgeries, will be collected and processed. Thereafter, the CSCs will be cultured and expanded from the RAA. The second screening will occur an average of 4 ± 1 months after CABG surgery, and will utilize a LVEF of < 40% assessed by cardiac MRI and/or the disk summation method [or Simpson's method] using echocardiography, for final enrollment.

* The preliminary eligibility criteria will utilize an EF < 40% measured by any of the following: cardiac imaging tests performed within 2 weeks prior to screening: echocardiography, gated SPECT and/or LV angiography.
* A maximum of 60 patients who satisfy the preliminary eligibility criteria will be enrolled in the preliminary phase of the study (i.e., will have RAA tissue harvested/cultured/expanded). Of these 60 patients, a maximum of 20 will be enrolled in the final phase of the study (i.e., will undergo CSC injections and subsequent follow-up).
* In this open-label study, a maximum of 20 patients will eventually receive intracoronary CSC transplantation. These patients will have nonviable myocardium/scar from prior MI and will undergo CABG for ICM.
* Enrollment of patients will be done in two stages: Stage A and stage B.
* In stage A, 9 consecutive patients will be enrolled in the treatment arm followed by 4 consecutive patients in the control arm. Stage A will enable us to perform an initial assessment of whether the process of harvesting, processing, and administering cardiac stem cells is associated with common/frequent short-term adverse effects.
* In stage B, patients will be randomized to the treated and control arms using a 2:3 ratio with a block size of 5 with a final variable block. As a result, the total number of both treated and control patients will be 20 each. More specifically, 11 treated and 16 control patients will make up stage B. To ensure that randomization can be done at the time of final enrollment, right atrial tissue will be harvested and cardiac stem cells will be grown from all patients who meet the enrollment criteria at the time of initial enrollment. If a patient is then randomized to the control arm, his/her cells will be discarded.
* Patients who satisfy the preliminary eligibility criteria will be enrolled and revascularized within few days (< 2 weeks) of enrollment.
* Patients will receive venous and/or arterial grafts as needed during CABG surgery. Nonviable myocardial segments will also be revascularized in order to enable subsequent intracoronary delivery of CSCs into the scarred region.
* During on-pump CABG surgery, patients will undergo resection of part of the RAA at the cannulation site (this is done routinely during CABG surgery). Resected RAA tissue (< 1 g) will be collected intra-operatively and handled as described in the preparation section.
* Cardiac catheterization (coronary angiography) for intracoronary injection of CSCs will be performed 4 ± 1 month after CABG surgery.

Worldwide, more than 500 patients have received intracoronary infusions of stem cells (derived from the bone marrow and peripheral blood). None of these patients have had any adverse events as a result of these infusions.

The overall objective of this project is to determine whether intracoronary delivery of CSCs can regenerate non-viable myocardial segments in patients with ICM. CSCs will be harvested from right atrial appendages (RAAs) of patients with ICM during surgical revascularization, cultured and expanded in vitro, and then transplanted back into the same patient.

The specific aims are:

1. To determine the feasibility of harvesting CSCs from RAAs of patients undergoing surgical revascularization, culturing and expanding them in vitro, and injecting them into patients via the intracoronary route
2. To determine the safety of intracoronary infusion of CSCs

In addition to these safety data, we hope to obtain initial evidence that CSC administration results in clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

* LVEF < 40% (by any imaging modality: echocardiography/SPECT/LV angiography)
* A history of Q-wave MI with a residual akinetic and nonviable scar (as evidenced by low-dose dobutamine stress echocardiogram and/or or thallium redistribution nuclear study for viability and/or an electrocardiogram)
* Patients scheduled for surgical revascularization within few days (< 2 weeks) of the initial screening

Exclusion Criteria:

* Age >75 by time of infusion
* Cardiogenic shock
* Severe co-morbidities (e.g., renal failure, liver failure)
* Mini-CABG procedures
* Pregnant/nursing women or women of child-bearing potential
* Inability to provide informed consent
* Diabetic Hgb A1c > 8.5%
* Patients with a history of hepatitis B, hepatitis C, and HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Monitoring adverse outcomes, death, sustained/symptomatic ventricular tachycardia, infection, bleeding, MI, stroke, peripheral embolism in the hospital after drug administration, in the first month after injection, and serially afterwards. | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bolli, MD, Principal Investigator — University of Louisville
Locations (1):
- Jewish Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chugh AR, Beache GM, Loughran JH, Mewton N, Elmore JB, Kajstura J, Pappas P, Tatooles A, Stoddard MF, Lima JA, Slaughter MS, Anversa P, Bolli R. Administration of cardiac stem cells in patients with ischemic cardiomyopathy: the SCIPIO trial: surgical aspects and interim analysis of myocardial function and viability by magnetic resonance. Circulation. 2012 Sep 11;126(11 Suppl 1):S54-64. doi: 10.1161/CIRCULATIONAHA.112.092627. PMID 22965994
- [Derived] Bolli R, Chugh AR, D'Amario D, Loughran JH, Stoddard MF, Ikram S, Beache GM, Wagner SG, Leri A, Hosoda T, Sanada F, Elmore JB, Goichberg P, Cappetta D, Solankhi NK, Fahsah I, Rokosh DG, Slaughter MS, Kajstura J, Anversa P. Retracted: Cardiac stem cells in patients with ischaemic cardiomyopathy (SCIPIO): initial results of a randomised phase 1 trial. Lancet. 2011 Nov 26;378(9806):1847-57. doi: 10.1016/S0140-6736(11)61590-0. Epub 2011 Nov 14. PMID 22088800 (Retraction: PMID 30894259 Lancet. 2019 Mar 16;393(10176):1084)